CLINICAL TRIAL: NCT04214301
Title: An Open-Label Preference Evaluation of BLI800
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLI800-491
Record Dates: First submitted 2019-12-27; First posted 2020-01-02 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BLI800 (Experimental): BLI800
  Interventions: Drug: BLI800

INTERVENTIONS:
Drug: BLI800 — BLI800 Bowel Preparation

SUMMARY:
The purpose of this study is to evaluate patient experience ratings of BLI800 in adult patients undergoing colonoscopy.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the patient satisfaction and preference of BLI800 in adult patients undergoing colonoscopy.

ELIGIBILITY:
Primary Inclusion Criteria:

* Male or female outpatients who are undergoing colonoscopy for a routinely accepted indication
* 18 to 85 years of age (inclusive)
* If female, and of child-bearing potential, is using an acceptable form of birth control
* Negative urine pregnancy test at screening, if applicable
* In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Primary Exclusion Criteria:

* Subjects with known or suspected ileus, severe ulcerative colitis, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon
* Subjects with ongoing severe, acute inflammatory bowel disease
* Subjects who had previous significant gastrointestinal surgeries
* Subjects with known severe renal, hepatic or cardiac insufficiency
* Subjects undergoing insulin therapy for any indication
* Subjects with impaired consciousness that predisposes them to pulmonary aspiration
* Subjects undergoing colonoscopy for foreign body removal and/or decompression

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mcgowan, MPH, Study Director — Braintree Laboratories, Inc.
Locations (2):
- United States (2):
  - Braintree Research Site 1, Great Neck, New York
  - Braintree Research Site 2, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BLI800
Started | 40
Completed | 38
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | BLI800
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Ease of Preparation Consumption
Description: Question: How easy or difficult was it to consume the study preparation?
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | BLI800
Number analyzed (Participants) | 38
Participants
  Very Difficult | 3
  Difficult | 5
  Tolerable | 15
  Easy | 7
  Very Easy | 8

2. Secondary Outcome: Preparation Compliance
Description: Question: Were you able to consume the entire preparation as instructed?
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | BLI800
Number analyzed (Participants) | 38
Participants
  Yes | 36
  No | 2

3. Secondary Outcome: Rating of Overall Experience
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | BLI800
Number analyzed (Participants) | 38
Participants
  Excellent | 9
  Good | 20
  Fair | 6
  Poor | 3
  Bad | 0

4. Secondary Outcome: Comparison to Prior Preparation
Description: How did this preparation experience compare to your prior experience?
Time Frame: 2 days
Population: Includes only those patients with a prior colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | BLI800
Number analyzed (Participants) | 22
Participants
  Worse | 2
  Same | 8
  Better | 12

5. Secondary Outcome: Willingness to Repeat Preparation
Description: Would you ask your doctor for this preparation again if you need another colonoscopy in the future?
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | BLI800
Number analyzed (Participants) | 38
Participants
  Yes | 30
  No | 8

6. Secondary Outcome: Refuse if Prescribed Again
Description: Would you refuse the same preparation again if it were to be prescribed to you in the future?
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | BLI800
Number analyzed (Participants) | 38
Participants
  Yes | 5
  No | 33

7. Secondary Outcome: Rating of Aftertaste
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | BLI800
Number analyzed (Participants) | 38
Participants
  Very Pleasant | 1
  Quite Pleasant | 6
  Neither Pleasant Nor Unpleasant | 15
  Quite Unpleasant | 11
  Very Unpleasant | 5

ADVERSE EVENTS:
Time Frame: 2 days
Groups:
- BLI800: BLI800 (SUPREP Bowel Prep Kit)
Arm/Group | BLI800
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 5/38
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI800 (N=38)
Bloating (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT04214301/Prot_SAP_000.pdf